CLINICAL TRIAL: NCT02696356
Title: A Phase 1, Open-Label, Multi-Center, Multi-Dose Study of Intradermal GRN-1201 in HLA-A*02 Subjects With Resected Stage IIb, IIc or III Melanoma
Brief Title: Phase 1 Study of GRN-1201 in HLA-A*02 Subjects With Resected Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BrightPath Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRN1201-001
Record Dates: First submitted 2016-02-03; First posted 2016-03-02 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Melanoma
Keywords: HLA-A*02
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): 0.1mg GRN-1201
  Interventions: Biological: GRN-1201
- Cohort 2 (Active Comparator): 1.0mg GRN-1201
  Interventions: Biological: GRN-1201
- Cohort 3 (Experimental): 3.0mg GRN-1201
  Interventions: Biological: GRN-1201

INTERVENTIONS:
Biological: GRN-1201 — GRN-1201 is a vaccine comprised of 4 peptides

SUMMARY:
This is a study of an investigational cancer vaccine called GRN-1201. Treatment with the GRN-1201 vaccine is a type of immunotherapy. The goal of immunotherapy is to stimulate the body's immune system (white blood cells) to attack cancer cells and kill them. GRN-1201 consists of 4 different peptides (small parts of proteins) that are expressed by melanoma cells. The intent of treatment with GRN-1201 is to increase your body's immune response to melanoma.

To further increase your body's immune response against tumor cells, the GRN-1201 vaccine will be mixed with Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF, also known as sargramostim). GM-CSF is a man-made protein that helps stimulate the immune system and increase the response against the tumor cells. This is a phase I study which means that this will be the first time GRN-1201 is given in combination with GM-CSF to humans. It will be tested in a small number of people to evaluate its safety, find a safe dose, and identify side effects. The safety of GRN-1201 will be tested at three different doses; the GM-CSF dose will remain the same.

DETAILED DESCRIPTION:
GRN-1201 is a novel HLA-A*02-restricted multiple-peptide, therapeutic cancer vaccine, being developed by GreenPeptide for the treatment of melanoma because it can induce immune responses against tumor associated antigens (TAAs), particularly cytotoxic T cell (CTL) responses. Granulocyte-macrophage-colony-stimulating-factor (GM-CSF) (Leukine®, SanofiAventis) will be administered in combination with GRN-1201 as an immuno-adjuvant

In contrast to advanced melanoma, treatment options in the adjuvant setting are limited. Surgical resection is the primary treatment of Stage IIb, IIc, and III melanoma patients. The rate of disease recurrence in patients with American Joint Committee on Cancer (AJCC) TNM Stage II (T2-4N0M0) and Stage III (TanyN+M0) disease ranges between 20 -60%, with 5-year overall survival between 45 - 70%. Thus, safe and effective treatment options to reduce the risk of recurrence are much needed. Considering their generally safe nature, peptide-based cancer vaccines would be ideal to address this unmet medical need. Patients with Stage IIb, IIc or III melanoma are, in general, healthy following local therapy. They are anticipated to maintain an immune system uncompromised by chemotherapy or disease burden. Further, they may have already developed immune response to TAAs targeted by GRN-1201, which may increase the probability of developing effective immune responses. It is conceivable that the combination of peptide vaccines with an immune checkpoint inhibitor, especially with a PD-1 pathway inhibitor, could enhance the efficacy of immunotherapy without increasing toxicity. Studies evaluating the combination of a melanoma vaccine with nivolumab in advanced melanoma [14] and resected high-risk metastatic melanoma patients [15] reported encouraging clinical outcome.

The pre-clinical data suggest that GRN-1201 may have anti-tumor activity in the adjuvant setting or may enhance activity of other drugs such as checkpoint inhibitors in the adjuvant or metastatic disease setting, by enhancing immune responses against TAAs.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥18 years of age (at the time consent is obtained);
* Provide written informed consent for study participation, approved by the appropriate institutional review board (IRB), and be willing and able to cooperate with all aspects of the protocol;
* Resected, histologically proven, cutaneous melanoma determined to be Stage IIb, IIc, or III; according to the American Joint Commission of Cancer Staging, 7th edition
* Human leukocyte antigen (HLA)-A*02+ by serology by an ASHI accredited laboratory;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0;
* Female subjects must have a negative serum human chorionic gonadotropic (hCG) test (pregnancy test not required for subjects with bilateral oophorectomy and/or hysterectomy or for those subjects who are >1 year post-menopausal); and
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 3 months after the last dose of study drug.

Exclusion Criteria:

* Inadequate hematologic or biologic function as determined by the following laboratory tests:
* Hemoglobin <10 g/dL,
* Platelet count <100,000/µL,
* Leukocyte count <3000/µL,
* Lymphocyte count <1000/µL,
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >2 × upper limit of normal (ULN),
* Total bilirubin >ULN: Subjects with Gilbert's syndrome are allowed if total bilirubin is <3.0 mg/dL and direct bilirubin is ≤ULN,
* Serum creatinine >ULN, or Prothrombin time (PT) or international normalized ratio (INR) >1.5 × ULN or activated partial thromboplastin time (aPTT) > 1.5 × ULN
* Greater than 3 months since melanoma resection;
* Have known fungal, bacterial, and/or viral infection, including human immunodeficiency virus (HIV) or hepatitis virus (B or C);
* Active immunosuppressive therapy associated with: Organ or allogeneic hematopoietic stem cell transplant, High-dose steroids, such as daily steroid doses in excess of 20 mg/day of prednisone (Note: Use of intra-articular or topical corticosteroids or eye drops containing corticosteroids is acceptable.), or Inhaled corticosteroids;
* Known history of autoimmune conditions including, but not limited to: rheumatoid arthritis, multiple sclerosis, lupus erythematosus, scleroderma, sarcoidosis, inflammatory bowel disease, idiopathic thrombocytopenia purpura, Graves' disease, or Hashimoto's thyroiditis;
* Current requirement for anti-coagulation therapy that prolongs PT or aPTT 7. History of prior malignancy except: Curatively treated non-melanoma skin cancer; Solid tumor treated curatively >5 years previously without evidence of recurrence; or History of other malignancy that in the Investigator's opinion would not affect the determination of study treatment effect (e.g., superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast);
* Non-healed wound;
* Prior adjuvant therapy for current melanoma diagnosis;
* History of any clinically significant cardiovascular disorder (i.e., symptoms above Class II per New York Heart Association [NYHA] Functional Classification);
* History of serious allergic reaction to yeast or yeast-derived products, including known or suspected hypersensitivity reaction to sargramostim;
* Pregnant, breastfeeding, or planning to become pregnant during the study;
* Received any other investigational therapy within 28 days of Day 1; or
* Any concurrent medical condition that, in the opinion of the Investigator, would complicate or compromise compliance with the study or the well-being of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Summary of number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0, | First dose through 16 weeks after last dose of study drug

SECONDARY OUTCOMES:
Immune response by gamma interferon ElliSpot assay | First dose through 16 weeks after last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Walter J Urba, MD, PhD, Principal Investigator — Providence Health and Services
Locations (4):
- United States (4):
  - The Christ Hospital Cancer Research, Cincinnati, Ohio
  - Providence Health and Services, Providence Portland Medical Center, Portland, Oregon
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No